CLINICAL TRIAL: NCT06889922
Title: The Effect of Low-Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) on Upper Extremity Spasticity and Spinal Excitability in Patients with Chronic Ischemic Stroke
Brief Title: The Effect of Low-Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Serhat Özdoğan, MD, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-PMR-Ozdogan
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-11

CONDITIONS: Spasticity, Post-Stroke
Keywords: Transcranial Magnetic Stimulation; Spasticity; Functional Recovery
MeSH Terms: conditions — Muscle Spasticity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): Patients received a total of 10 sessions active rTMS on M1 region of the non-lesional hemisphere. TMS coil was initially placed tangentially to the scalp over the presumed motor cortex area. The motor hotspot is defined as the location where the lowest stimulus intensity consistently produces a significant motor-evoked potentials (MEP) in the first dorsal interosseous muscle. Once the hotspot was identified, the resting motor threshold (rMT) was determined as the lowest single pulse TMS intensity required to produce a MEP amplitude larger than 50 mV in more than 5 out of 10 trials from the first dorsal interosseous muscle. 1200 pulses at 90% of the rMT were delivered to the hotspot of the first dorsal interosseous muscle in the contralesional hemisphere. A routine physical therapy and rehabilitation program, including range of motion exercises for the upper extremity, neurophysiological exercises, and occupational therapy, was applied to patients within 30 min after TMS sessions.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Patients received a total of 10 sessions sham rTMS on M1 region of the non-lesional hemisphere. However, a sham coil was used for stimulation, thus no actual stimulation was administered to the patients. Instead, the sham coil produced a sensation resembling real stimulation, with sounds and sensations on the scalp that simulated the feeling of active stimulation. A routine physical therapy and rehabilitation program, including range of motion exercises for the upper extremity, neurophysiological exercises, and occupational therapy, was applied to patients within 30 min after TMS sessions.
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Magstim Rapid2 Magnetic Stimulator (Magstim, Whitland Dyfed, UK), 70 mm Figure-of-eight Coil
  Arms: Active rTMS
Device: Transcranial Magnetic Stimulation Sham — Magstim Rapid2 Magnetic Stimulator (Magstim, Whitland Dyfed, UK), 70 mm Figure-of-eight Sham Coil
  Arms: Sham rTMS

SUMMARY:
In this study, we aimed to demonstrate the effects of 1 Hz rTMS applied to the contralesional hemisphere on upper extremity spasticity, spinal excitability, and additionally on motor recovery in stroke patients in the chronic phase with clinically and electrophysiological parameters (Hmax/Mmax).

DETAILED DESCRIPTION:
Post-stroke spasticity is a common complication that can severely impact daily living activities, causing pain and hygiene challenges for a significant number of patients. Spasticity is a clinical condition that arises as a result of abnormal or hyperexcitable spinal reflexes, and the excitability of the spinal stretch reflex is regulated through supraspinal descending pathways such as the Dorsal Reticulospinal tract, Medial Reticulospinal tract, and Vestibulospinal tract. The treatment of spasticity can be categorized into non-pharmacological, pharmacological, and surgical approaches. Pharmacological options include Baclofen, Tizanidine, Dantrolene, and Botulinum toxin injections. However, these treatments may cause side effects such as sedation, cognitive impairment, and muscle weakness. The application of Repetetive Transcranial Magnetic Stimulation (rTMS) is based on the hypothesis that neuromodulation, achieved by inhibiting the contralesional hemisphere with 1 Hz stimulation or facilitating the ipsilesional hemisphere with stimulation above 1 Hz, can normalize interhemispheric inhibition.The search for alternative effective treatments and the aim to minimize undesirable side effects have led to a significant rise in studies exploring the effects of rTMS on spasticity in recent years.

Our study is a randomized, double-blind, sham-controlled clinical trial. According to the statistical analysis 20 patients who were registered at Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital between July 2021 and May 2022 and met the study criteria were included. Patients were divided into two groups using a computer-based randomization program: a 1 Hz rTMS group (n=10) and a sham group (n=10). The researcher conducting the clinical assessments was blinded to the group assignments of the patients. Furthermore, the patients themselves were unaware of which group they had been assigned to. Active stimulation was applied to the M1 region of the non-lesional hemisphere using a 70-mm figure-eight coil, while the sham group received the same protocol with a sham coil that visually resembled the active coil. The coil was initially placed tangentially over the presumed motor cortex, and the motor hotspot was identified by applying single pulses at different positions until the lowest intensity produced a significant motor-evoked potential (MEP) in the first dorsal interosseous muscle. The resting motor threshold (rMT) was then determined as the lowest intensity to produce an MEP amplitude larger than 50 mV in more than 5 out of 10 trials. In the active treatment group, 1200 pulses at 90% of rMT were delivered to the hotspot of the first dorsal interosseous muscle in the contralesional hemisphere across 10 sessions over two weeks, while the sham group received sham stimulation. Safety protocols were followed, and both groups underwent physical therapy, including upper extremity exercises and occupational therapy, within 30 minutes after each TMS session.

Clinical evaluations were conducted three times for each patient: Baseline (before treatment), 2nd week (at the and of treatment), and 6th week.

ELIGIBILITY:
Inclusion Criteria:

* Having a lesion in a single hemisphere confirmed by MRI,
* At least 6 months and at most 2 years having passed since the stroke,
* Spasticity in wrist flexors and finger flexors at levels 1+, 2, or 3 according to the modified Ashworth scale,
* Being between 18-75 years old,
* Having a Mini-Mental Test score of ≥ 24,
* If using antispastic medication, no change in medication dosage in the last month.

Exclusion Criteria:

* History of epilepsy, dementia, cognitive impairment, or neurodegenerative disease,
* Having a metallic materials in the area to be stimulated (such as a cochlear implant, brain pacemaker, or drug pump),
* Alcoholism,
* Pregnancy,
* Severe and newly decompensated heart failure,
* Using medications that lower the seizure threshold.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | Baseline (before treatment), 2nd week (at the end of treatment), 6th week
  The Modified Ashworth Scale (MAS) is an updated version of the original Ashworth Scale, designed to assess spasticity in patients with central nervous system disease. It measures the increase in muscle tone, assigning a spasticity grade on a 0-4 ordinal scale. 0: no increase in muscle tone, 1: minimal resistance at the end of the range of motion, 1+: slight increase in muscle tone less than half of the ROM, 2: increase in muscle tone through most of the ROM, 3: considerable increase in muscle tone, passive movement difficult, 4: affected parts rigid.
Electromyography - H-reflex (Hmax/Mmax) | Baseline (before treatment), 2nd week (at the end of treatment), 6th week
  The H reflex is the electrophysiological analogue of the stretch reflex. An increase in the amplitude of the H reflex is an indicator of spinal excitability. The peak-to-peak amplitude of the highest H reflex obtained from the flexor carpi radialis muscle (Hmax) is expressed as the ratio of the peak-to-peak amplitude of the maximum M response (Mmax) to Hmax (Hmax/Mmax). A higher Hmax/Mmax ratio obtained from the flexor carpi radialis muscle indicates reduced voluntary motor activity and increased reflex excitability.

SECONDARY OUTCOMES:
Fugl-Meyer Upper Extremity Motor Assessment Scale | Baseline (before treatment), 2nd week (at the end of treatment), 6th week
  Fugl-Meyer Upper Extremity Motor Assessment Scale used to determine the severity of motor impairment and to evaluate the effectiveness of therapeutic interventions. The assessment is conducted in 9 different categories. These are: reflex activity, flexor synergy, extensor synergy, movements performed with a combination of flexor and extensor synergies, movements performed with minimal or without synergy, normal reflex activity (only for those who score full points on step 5), wrist, hand, coordination and speed. Scoring is determined through direct observation of the patient's performance. Each item on the scale is scored using a 3-point ordinal scale based on the ability to complete the task, where 0 indicates "cannot perform," 1 indicates "performs partially," and 2 indicates "performs fully."

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yalçın, Prof, MD, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No